CLINICAL TRIAL: NCT06492187
Title: Triage Survey for Infectious Disease Eligibility (SWIFT-ID-101)
Brief Title: Triage Survey for Infectious Disease Eligibility
Status: Recruiting | Type: Observational
Sponsor: Brooklyn Clinical Research (Network)
Responsible Party: Sponsor
Other Study IDs: SWIFT-ID-101
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Vaccination; Infection; HIV-1-infection; Infectious Disease
MeSH Terms: conditions — Infections; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SWIFT-ID-101 is a single site survey study designed to assess potential participants' eligibility to screen for industry-sponsored clinical trials for diagnosis, treatment, or prevention of infectious diseases such as in the areas of HIV, vaccines, and other infectious-diseases areas. A physician will oversee the informed consent process, after which participants will be surveyed on demographics, medical/surgical history, physical examination, comorbidities, and any current symptoms. Informed consent will be done electronically (preferable) or on paper. Informed consent may be done in-person or remotely, depending on patient preference. Information related to HIV, hepatitis B and C, other infectious diseases, or substance use disorder will also be obtained if applicable. Site staff may collect vital signs, fingerpick testing, urine drug screens, blood draws, EKG, and pregnancy tests. Some testing may be recommended in a fasting condition. A doctor will review medical history and results of the above evaluations with the participant to determine study suitability via clinical interview. The doctor may reach out to the patient's current treating physicians, other providers, and pharmacies to determine eligibility for clinical trials. A follow-up phone call may be needed to discuss testing results and/or trial eligibility. If a participant is deemed eligible for future trials and if the participant remains interested, counseling on contraception requirements for trials will be discussed.

ELIGIBILITY:
Inclusion Criteria:

- 1. Participant or Legally Authorized Representative has signed an ICF prior to study-specific procedures being performed.

2. Participant is at least 18 years old.

Exclusion Criteria:

1. Participants are pregnant, breast-feeding, or planning to become pregnant.
2. History of a clinically significant illness which in the investigator's opinion may impact participant safety or the ability to analyze study results or makes them unsuitable for the study for another reason.
3. Current or recent moderate or severe substance use disorder impacting their ability to follow study related procedures.
4. Reported history of coagulopathy or bleeding disorder considered a contraindication to phlebotomy.
5. Any condition that in the investigator's opinion makes a participant unsuitable for the clinical trial study.
6. Currently employed by Swift Clinical Research Group, Inc. or any of its subsidiaries, including Brooklyn Clinical Research, or a first-degree relative of an employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total of the program, we anticipate 10,000 participants of any sex, gender, age 18+, who have expressed interest in participating in a clinical trial of an investigational product such as device or drug, for indications in infectious diseases related therapeutic areas will be screened for clinical appropriateness for a study trial.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2029-01-28 (Estimated); Study Completion 2029-01-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants interested in clinical research | 5 years
  Number of participants for whom an industry-sponsored clinical research clinical research is clinically appropriate for HIV, vaccines, and other infectious diseases

SECONDARY OUTCOMES:
Clinical Trial Enrollment | 5 years
  Proportion of the clinical trial seeking population who enroll in industry-sponsored studies in infectious diseases therapeutic area.

OTHER OUTCOMES:
Disqualifying conditions | 5 years
  Prevalence of disqualifying comorbid conditions that prevent screening or enrollment in industry-sponsored clinical research for HIV, vaccines, and other infectious diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooklyn Clinical Research, Brooklyn, New York, United States